CLINICAL TRIAL: NCT00261872
Title: Treatment of Patients With Alcoholism and Attention Deficit Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060004; 06-AA-0004
Record Dates: First submitted 2005-12-03; First posted 2005-12-05 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-04-09

CONDITIONS: Alcoholism; Attention Deficit Disorder
Keywords: Alcoholism; Attention Deficit Disorder; ADHD
MeSH Terms: conditions — Alcoholism; Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

INTERVENTIONS:
Drug: Methylphenidate

SUMMARY:
This study of persons with both alcoholism and ADHD will determine whether adding the drug methylphenidate to a standard treatment program will decrease alcohol use. In approximately half of patients with ADHD, symptoms persist into adulthood, and the untreated condition is associated with a significantly increased incidence of substance use disorder. Also, more than one-third of adults with substance use disorder have symptoms of ADHD. This study will evaluate the effectiveness of adding methylphenidate to a standard alcohol treatment program in improving patients' treatment compliance and decreasing adverse consequences of drinking, as well as monitoring their attention deficit/hyperactivity symptoms,

People 21 to 65 years of age with alcoholism and attention deficit hyperactivity disorder (ADHD) may be eligible for this study.

Participants are randomly assigned to receive either slow-release methylphenidate (an approved medication for ADHD) or placebo. All subjects participate in NIAAA's alcohol treatment program, which includes a standardized 12-week behavioral therapy course and treatment with naltrexone, a medication to prevent relapse. Patients are assessed once a week with the standard NIAAA treatment evaluation battery, including:

* Timeline Followback: A validated self-report method to assess a person's drinking over a defined interval in time
* Addiction Severity Index: A validated interview that measures problem severity in seven areas related to drug and alcohol abuse
* Biomarkers for alcohol abuse
* Conners Adult ADHD Rating Scale (a rating scale for ADHD symptoms and severity)

DETAILED DESCRIPTION:
Background: Several pharmacological therapies for relapse prevention in alcoholism have now been documented for efficacy. A key issue that has emerged is the role of patient compliance with medication in mediating efficacy. Psychological traits common among alcoholics interact with treatment compliance. Thus, a considerable proportion of alcoholics, e.g. more than one third of treatment seeking populations, display signs and symptoms of adult ADHD. The impaired ability for long term planning and sustained goal-oriented behaviors in this group is likely to impair compliance with pharmacological treatment, thus reducing its potential beneficial effects.

Well documented pharmacological treatments are also available for ADHD. Among these, methylphenidate has a strong documentation, and has been demonstrated to be as efficacious in adult ADHD as in the childhood condition. A recently introduced slow release preparation of methylphenidate appears to offer considerable advantages, in that it eliminates most of the abuse potential, and allows once daily administration.

Aims: The aim of this study is to evaluate whether addition of methylphenidate to a state of the art treatment program for alcohol dependence will improve clinically relevant treatment outcomes such as validated measures of alcohol drinking.

Methods: The hypothesis will be addressed in a 12 week randomized, placebo controlled double blind add-on trial. Participation will be offered to subjects with alcohol dependence, aged 21-65 years, who enter the NIAAA alcohol treatment program, do not have any severe psychiatric or physical morbidity, and meet criteria for adult ADHD. All patients who are included will be given a standardized state of the art 12 week behavioral treatment package, as well as naltexone, an approved medication for relapse prevention. In addition subjects will be randomized to slow release methylphenidate or corresponding placebo. Patients will be evaluated upon weekly visits using the standard NIAAA treatment evaluation battery TLFB, ASI, biomarkers, as well as the established CAARS rating scale for attention deficit / hyperactivity. Primary outcome will be measures of drinking obtained by the TLFB methodology. Secondary outcomes will measures of attention deficit and hyperactivity, as measured by the CAARS scores.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 21 or older.

DSM-IV diagnosis of alcohol dependence or alcohol abuse on SCID, and alcohol problems as primary complaint among SUD:s

DSM-IV diagnosis of ADHD on SCID, confirmed by CAARS-INV

EXCLUSION CRITERIA:

General exclusion criteria for the NIAAA intramural treatment program:

1. People who present with complicated medical problems requiring intensive medical or diagnostic management, such as hypertensive emergency, serious GI bleeding, major organ or body system dysfunction such as decompensated liver disease, renal failure, myocardial ischemia, congestive heart failure or cerebrovascular disease, major endocrine problems such as uncontrolled diabetes, pancreatic or thyroid disease.
2. People who are infected with the Human Immunodeficiency Virus (HIV).
3. Serious neuro-psychiatric conditions which impair judgment or cognitive function to an extent that precludes them from providing informed consent or complying with treatment, such as psychotic illness or severe dementia (incompetent individuals).
4. People who are unlikely or unable to complete the treatment program because they become or are likely to be incarcerated while on the protocol.
5. People who are required to receive treatment by a court of law or who are involuntarily committed to treatment.
6. People with uncontrolled hypertension
7. People with a history of withdrawal seizures

Study specific exlusion criteria:

1. Pregnancy or lactation (negative pregnancy test required)
2. Use of psychotropic medication (antidepressant, lithium, antipsychotic, anxiolytic, antiepileptic) within last 4 weeks, except when given within the program as part of medically supervised withdrawal. Use of these medications constitutes prima facie evidence of general exclusion category 3 (above). Persons identified with psychiatric conditions deemed exclusionary will be referred to community resources for inpatient or outpatient treatment as indicated. Persons with acute psychiatric emergencies (e.g. bipolar disorder, manic phase, significant depressive symptoms, or active suicidal ideation) will be referred for immediate care to ensure safety and stabilization; such actions will be appropriately documented.
3. Past DSM-IV diagnosis of dependence (but not abuse, or reported occasional use of) drugs of abuse other than alcohol.
4. Present DSM-IV diagnosis (but not sporadic use) of dependence on any central stimulant
5. Present use of guanethidine or yohimbine
6. Contraindications / warnings for naltrexone (in addition to those included in the general exclusion criteria):

1. known supersensitivity to the drug

2. acute hepatitis (any transaminase great than 3 x upper normal interval limit)

3. ongoing (within last month) use of opid analgesics, or illicit opiates

7. Contraindications / warnings for methylphenidate (in addition to those included in the general exclusion criteria):

1. known supersensitivity to the drug
2. marked anxiety, tension or agitation, since the drug may aggravate these symptoms
3. glaucoma
4. motor tics, or family history or diagnosis of Tourettes syndrome
5. history of seizures
6. hypertension, or known disease which can be aggravated by an elevation of blood pressure or increased pulse rate

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-12-01; Study Completion 2007-04-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] COMBINE Study Research Group. Testing combined pharmacotherapies and behavioral interventions for alcohol dependence (the COMBINE study): a pilot feasibility study. Alcohol Clin Exp Res. 2003 Jul;27(7):1123-31. doi: 10.1097/01.ALC.0000078020.92938.0B. PMID 12878918